CLINICAL TRIAL: NCT01088893
Title: A Randomized Study of mTOR Inhibition by RAD001 (Everolimus) in Invasive Breast Cancer Patients After Pre-operative Use of Anthracycline and/or Taxane-based Chemotherapy
Brief Title: Everolimus in Breast Cancer Patients After Pre-operative Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Organisation for Oncology and Translational Research (Other)
Responsible Party: Senior Manager, OOTR
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OOTR-N006
Record Dates: First submitted 2009-08-11; First posted 2010-03-17 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-05

CONDITIONS: Breast Neoplasms
Keywords: everolimus; neoadjuvant; m-TOR inhibitor
MeSH Terms: conditions — Breast Neoplasms | interventions — Everolimus

ARMS (2):
- observation (No Intervention)
- Everolimus (Experimental)
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — 10mg/d) for three weeks 1 week after completion of neoadjvuant treatment and before surgery
  Arms: Everolimus

SUMMARY:
This is a randomized controlled pilot study investigating signals involved in drug resistance to chemotherapy.

Patient will be randomized to undergo observation or to receive Everolimus after completion of neoadjvuant treatment (anthracycline and/or taxane-based) and before surgery. The patients will be monitored for efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥ 18 years;
* Histologically and/or cytologically confirmed invasive ductal or lobular breast cancer;
* Tumor of 3 cm or greater at time of diagnosis
* Measurable primary tumor after neoadjuvant treatment before randomization
* No prior chemotherapy for breast cancer;
* ECOG performance status ≤1 or Karnofsky performace status ≥ 70%
* Adequate liver/renal function
* Able to swallow whole tablets.
* Able to give written informed consent
* Able to follow prescription instructions reasonably well

Exclusion Criteria:

* Male patient
* Prior history of other malignancy within 5 years of study entry, aside from contralateral breast carcinoma, appropriately treated cervical carcinoma in situ, or adequately treated basal or squamous cell carcinoma of the skin
* Distant metastasis, including skin involvement beyond the breast area
* Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that would impart, in the judgment of the investigator, excess risk associated with study participation or study drug administration, or which, in the judgment of the investigator, would make the patient inappropriate for entry into this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-11; Primary Completion 2012-12 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
measure change of biomarkers in pre- and post- surgery samples | baseline and 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Unimed Medical Institute, Hong Kong, China